CLINICAL TRIAL: NCT04255186
Title: Treatment Using 448 kHz Capacitive Resistive Monopolar Radiofrequency in Patients With Subacromial Syndrome. A Randomised Controlled Trial.
Brief Title: Treatment Using 448 kHz CRMRF in Subacromial Syndrome.
Acronym: CRMRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Hospital General Nuestra Señora del Prado (Other); Castilla-La Mancha Health Service (Other); Indiba S.A. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 448 kHz CRMRF UCLM
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Shoulder Impingement Syndrome; Subacromial Impingement Syndrome
Keywords: shoulder pain; shoulder impingement syndrome; radiofrequency treatment; electrophysical agents
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thermal CRMRF (Experimental): 9 sessions in 3 week of Thermal CRMRF: The power of the RFCR equipment in this intervention will be 35 VA in capacitive method (10% of the maximum power of the equipment) and 30 W in the resistive method (15% of the maximum power of the equipment) in 3 week (3 sessions a week on alternate days) + 15 sessions in 3 week of exercise protocol (5 sessiones a week).
  In Thermal CRMRF it will be necessary to adapt to the patient's thermal sensitivity
  Interventions: Device: Thermal 448 kHz Capacitive Resistive Monopolar Radiofrequency
- Subthermal CRMRF (Experimental): 9 sessions in 3 week of Subthermal CRMRF: The power of the RFCR equipment in this intervention will be 7 VA in capacitive method (2% of the maximum power of the equipment) and 4 W in the resistive method (2% of the maximum power of the equipment) in 3 week (3 sessions a week on alternate days) + 15 sessions in 3 week of exercise protocol (5 sessions a week).
  Interventions: Device: Subthermal 448 kHz Capacitive Resistive Monopolar Radiofrequency
- Sham CRMRF (Sham Comparator): 9 sessions in 3 week of sham stimulation: The application will be carried out in the same way as in the experimental groups, but in this case the manufacturer will introduce a simulated stimulation protocol so that the device does not emit current + 15 sessions in 3 week of exercise protocol (5 sessiones a week).
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Thermal 448 kHz Capacitive Resistive Monopolar Radiofrequency — Thermal Application of 448 kHz monopolar radio frequency in capacitive and resistive method
  Other Names: CRMRF
  Arms: Thermal CRMRF
Device: Subthermal 448 kHz Capacitive Resistive Monopolar Radiofrequency — Subthermal Application of 448 kHz monopolar radio frequency in capacitive and resistive method
  Arms: Subthermal CRMRF
Device: Sham stimulation — a simulated stimulation protocol so that the device does not emit current
  Arms: Sham CRMRF

SUMMARY:
The purpose of this study is to assess the effectiveness of 448 kHz capacitive resistive monopolar radiofrequency in the treatment of subacromial syndrome.

DETAILED DESCRIPTION:
Shoulder pain has a high prevalence in our society, several studies estimate an annual prevalence between 5% and 47%. It is one of the main causes of musculoskeletal pain, particularly in third place, after the low back pain and neck pain.

Symptoms of pathologies of subacromial syndrome, where, regardless of origin, pain is the number one symptom for the patient, which emanates functional impairment and the impact on quality of life.

Among the non-pharmacological treatments of subacromial syndrome, a systematic review concludes that the first line of intervention should be a therapeutic exercise program. In many cases, this is usually accompanied by the application of electrophysical agents (short wave, laser, etc.). A recent study has shown that the application of Short Wave Radio Frequency improved pain in people with subacromial syndrome. The current frequency that is applied in the short wave is 27.12 MHz, however, there are other relatively new forms of radiofrequency in which a frequency less than 1 MHz is used. These are beginning to be used in clinical practice and recently have shown positive results related to pain and functionality of musculoskeletal pathologies such as knee osteoarthritis. In these two clinical trials, what is called Resistive Capacitive Monopolar Radio Frequency (RFCR) was used, the frequency of which was 448 KHz and 485KHz respectively, much lower than the frequency used in Shortwave. The RFCR has a potential advantage since it is applied with electrodes directly on the skin and is not transmitted in the air unlike the Short Wave.

Based on the few clinical trials in people with pathology and the physiological effects evidenced in healthy people and in vitro preclinical studies, it is considered pertinent to carry out the present investigation.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 70 years years old with diagnosis of subacromial syndrome
* Visual Analogue Scale (VAS) less than or equal to 7.
* Positive Neer and Hawkins test.

Exclusion Criteria:

* Clinical examination compatible with complete rotator cuff tear (Drop-arm positive test)
* Fibromyalgia
* Adhesive capsulitis
* Be receiving physiotherapeutic treatment or have received it previously for this pathology one month before the start of treatment.
* Patients with alterations of thermal sensitivity.
* Derived from the absolute and relative contraindications of CRMRF:
* Pacemaker
* Thrombophlebitis
* Pregnancy
* Skin disorders (recent wounds or burns)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Baseline
  minimun 0 - maximun10. Higher scores mean a worse outcome
Visual Analogue Scale | After 3 weeks
  minimun 0 - maximun10. Higher scores mean a worse outcome
Visual Analogue Scale | 1 month after the end of the intervention
  minimun 0 - maximun10. Higher scores mean a worse outcome
Visual Analogue Scale | 3 months after the end of the intervention
  minimun 0 - maximun10. Higher scores mean a worse outcome
SPADI | Baseline
  Shoulder Pain and Disabilty Index
SPADI | After 3 weeks
  Shoulder Pain and Disabilty Index
SPADI | 1 month after the end of the intervention
  Shoulder Pain and Disabilty Index
SPADI | 3 months after the end of the intervention
  Shoulder Pain and Disabilty Index

SECONDARY OUTCOMES:
Quick DASH | Baseline
  Abbreviated
Quick DASH | After 3 weeks
  Abbreviated
Quick DASH | 1 month after the end of the intervention
  Abbreviated
Quick DASH | 3 months after the end of the intervention
  Abbreviated
PPT | Baseline
  Pressure Pain Threshold in subacromial area
PPT | After 3 weeks
  Pressure Pain Threshold in subacromial area
European Quality ol life - 5 dimensions (EQ-5D) | Baseline
  Higher scores mean a better outcome
European Quality ol life - 5 dimensions (EQ-5D) | After 3 weeks
  Higher scores mean a better outcome
European Quality ol life - 5 dimensions (EQ-5D) | 1 month after the end of the intervention
  Higher scores mean a better outcome
European Quality ol life - 5 dimensions (EQ-5D) | 3 months after the end of the intervention
  Higher scores mean a better outcome

OTHER OUTCOMES:
Medication intake | Baseline
  Analgesic ladder for chronic pain. Higher scores mean a worse outcome
Medication intake | After 3 weeks
  Analgesic ladder for chronic pain. Higher scores mean a worse outcome
Medication intake | 1 month after the end of the intervention
  Analgesic ladder for chronic pain. Higher scores mean a worse outcome
Medication intake | 3 months after the end of the intervention
  Analgesic ladder for chronic pain. Higher scores mean a worse outcome
Blinding assesment | After three weeks
  The patient, the external evaluator, the therapist who applies radiofrequency and the kinesitherapist physiotherapist will be asked about the patient's group of belonging.
Blinding assesment | 3 months after the end of the intervention
  The patient, the external evaluator, the therapist who applies radiofrequency and the kinesitherapist physiotherapist will be asked about the patient's group of belonging.
Total number of sessions of the exercise protocol for discharge | 3 months after the end of the intervention
  After the first 3 weeks, if the patient has not met the criteria for discharge, more sessions will continue performing the same exercise protocol according to medical criteria. This total number of sessions will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Avendaño-Coy, PhD, Principal Investigator — Castilla La Mancha University; Javier Aceituno-Gómez, PhD, Principal Investigator — Castilla-La Mancha Health Service
Locations (1):
- Hospital General Universitario Nuestra Señora del Prado, Talavera de la Reina, Toledo, Spain